CLINICAL TRIAL: NCT03586921
Title: Group Therapy in Primary Care for Women With Depression or Anxiety in Petropolis
Brief Title: Primary Care Group Therapy for Depression/Anxiety for Women in Petropolis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rio de Janeiro State University (Other)
Responsible Party: Principal Investigator, Rosely Sichieri, Associate Professor, Rio de Janeiro State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DEP-ANX_PETROPOLIS
Record Dates: First submitted 2018-03-21; First posted 2018-07-16 (Actual); Last update posted 2018-07-16 (Actual); Status verified 2018-07

CONDITIONS: Depression; Anxiety Disorders
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: All patients received enhanced primary care, which included: (1) The nurses and doctors from the Family Health Teams were trained by Matrix team mental health professionals on clinical aspects of depression and anxiety, including diagnosis, appropriate medication interventions, psycho-education, and cognitive and problem solving therapy. (2) Given the high co-occurrence of anxiety and depression, the intervention was modified from the depression-only Chile model to emphasize co-occurring anxiety and depression in diagnoses, appropriate prescription of anxiolytics and antidepressants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced usual care + group intervention (Experimental): Intervention patients received enhanced primary care plus a 9-session group intervention. The intervention included two psycho-educational sessions with information about depression and anxiety disorders, two sessions on the development of pleasant activities including relaxation exercises, two sessions on solving problems therapy, one session on the problem of overcoming negative thoughts and emotions, one session on relapse prevention, and a final closure and review session which included a small party. The patients from the intervention arm also received additional outreach from the Family Health Teams, including home delivery of psychotropic medication when needed and active outreach and engagement by community workers if patients missed group sessions.
  Interventions: Behavioral: Psychosocial Group Intervention
- Enhanced Usual Care (Active Comparator): All patients received enhanced primary care: (1) Nurses and doctors from the Family Health Teams were trained by Matrix team mental health professionals on clinical aspects of depression and anxiety. (2) Given the high co-occurrence of anxiety and depression, the intervention was modified from the depression-only Chile model to emphasize co-occurring anxiety and depression in diagnoses, appropriate prescription of anxiolytics and antidepressants. (3) All providers received weekly group or individual consultation with a Matrix team mental health professional, either psychiatrist or psychologist. An qualitative study of participating Petrópolis Family Health Programme doctors and nurses demonstrated their satisfaction with the training.
  Interventions: Other: Enhanced Usual Care

INTERVENTIONS:
Behavioral: Psychosocial Group Intervention — The intervention included two psycho-educational sessions with information about depression and anxiety disorders, two sessions on the development of pleasant activities including relaxation exercises, two sessions on solving problems therapy, one session on the problem of overcoming negative thoughts and emotions, one session on relapse prevention, and a final closure and review session which included a small party.
  Arms: Enhanced usual care + group intervention
Other: Enhanced Usual Care — All patients received enhanced primary care: (1) Nurses and doctors from the Family Health Teams were trained by Matrix team mental health professionals on clinical aspects of depression and anxiety. (2) Given the high co-occurrence of anxiety and depression, the intervention was modified from the depression-only Chile model to emphasize co-occurring anxiety and depression in diagnoses, appropriate prescription of anxiolytics and antidepressants. (3) All providers received weekly group or individual consultation with a Matrix team mental health professional, either psychiatrist or psychologist. An qualitative study of participating Petrópolis Family Health Programme doctors and nurses demonstrated their satisfaction with the training.
  Arms: Enhanced Usual Care

SUMMARY:
This is a randomized controlled trial comparing two groups: 1) Enhanced usual care and 2) Enhanced usual care plus group psychological intervention. In both groups a "stepped care" approach was used to the management of anxiety and depression among women seen in primary care.

DETAILED DESCRIPTION:
All patients received enhanced primary care, which included: (1) The nurses and doctors from the Family Health Teams were trained by Matrix team mental health professionals on clinical aspects of depression and anxiety, including diagnosis, appropriate medication interventions, psycho-education, and cognitive and problem solving therapy. (2) Given the high co-occurrence of anxiety and depression, the intervention was modified from the depression-only Chile model to emphasize co-occurring anxiety and depression in diagnoses, appropriate prescription of anxiolytics and antidepressants. (3) All providers received weekly group or individual consultation with a Matrix team mental health professional, either psychiatrist or psychologist. An qualitative study of participating Petrópolis Family Health Programme doctors and nurses demonstrated their satisfaction with the training.

Patients in the intervention arm received enhanced primary care plus a 9-session group intervention (seven sessions weekly then two sessions every 15 days). The intervention included two psycho-educational sessions with information about depression and anxiety disorders, two sessions on the development of pleasant activities including relaxation exercises, two sessions on solving problems therapy, one session on the problem of overcoming negative thoughts and emotions, one session on relapse prevention, and a final closure and review session which included a small party. The patients from the intervention arm also received additional outreach from the Family Health Teams, including home delivery of psychotropic medication when needed and active outreach and engagement by community workers if patients missed group sessions.

ELIGIBILITY:
Inclusion Criteria:

* female patients who came to the primary care unit for any type of consultation for themselves (e.g., not for a child).
* General Health Questionnaire positive screen (>5 at two time points)
* positive diagnosis of depression or anxiety per the Mini Mental State Examination.

Exclusion Criteria:

* diagnosis of bipolar disorder, mania, severe suicidal ideation
* cognitive impairment that would limit their ability to consent or take part in the study. -pregnant.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Since this is a study of depression in women, we included only those who identify as women.
Enrollment: 340 (Actual)
Dates: Start 2006-05-19 (Actual); Primary Completion 2007-09-25 (Actual); Study Completion 2008-01-15 (Actual)

PRIMARY OUTCOMES:
Depression (Beck Depression Inventory) | Change in depression 4 months post intervention
  Depression measured by the Beck Depression Inventory
Depression (Beck Depression Inventory) | Change in depression 8 months post intervention
  Depression measured by the Beck Depression Inventory

SECONDARY OUTCOMES:
Anxiety (Beck Anxiety Inventory) | 4 months post intervention
  Anxiety as measured by the Beck Anxiety Inventory
Anxiety (Beck Anxiety Inventory) | 8 months post intervention
  Anxiety as measured by the Beck Anxiety Inventory
Quality of Life (World Health Organization Quality of Life Assessment, Brief Version) | 4 months and 8 months post intervention
  QoL as measured by the World Health Organization Quality of Life Assessment, Brief Version
Quality of Life (World Health Organization Quality of Life Assessment, Brief Version) | 4 months post intervention
  QoL as measured by the World Health Organization Quality of Life Assessment, Brief Version
Quality of Life (World Health Organization Quality of Life Assessment, Brief Version) | 8 months post intervention
  QoL as measured by the World Health Organization Quality of Life Assessment, Brief Version

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-12): https://cdn.clinicaltrials.gov/large-docs/21/NCT03586921/Prot_SAP_000.pdf